CLINICAL TRIAL: NCT04507932
Title: Characterizing Inflammatory Bowel Disease With 68Ga-FAPI PET/CT
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PekingUMCHFAPIIBD
Record Dates: First submitted 2020-08-07; First posted 2020-08-11 (Actual); Last update posted 2021-01-26 (Actual); Status verified 2021-01

CONDITIONS: Inflammatory Bowel Disease
MeSH Terms: conditions — Inflammatory Bowel Diseases | interventions — 68Ga-FAPI

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 68Ga-FAPI, PET/CT (Experimental): Inject 68Ga-FAPI and then perform PET/CT scan.
  Interventions: Drug: 68Ga-FAPI

INTERVENTIONS:
Drug: 68Ga-FAPI — Intravenous injection of one dosage of 74-148 MBq (2-4 mCi) 68Ga-FAPI. Tracer doses of 68Ga-FAPI will be used to image lesions of inflammatory bowel disease by PET/CT.
  Other Names: 68Ga-fibroblast activating protein inhibitors

SUMMARY:
68Ga-FAPI has been developed as a tumor-targeting agent as fibroblast activation protein is overexpressed in cancer-associated fibroblasts and some inflammation,such as inflammatory bowel disease. And it might be more sensitive than FDG in detecting a certain type of inflammations according to our preliminary research. Thus this prospective study is going to investigate whether 68Ga-FAPI PET/CT may be superior for diagnosis, therapy response assessment and follow-up of inflammatory bowel disease than 18F-FDG PET/CT.

DETAILED DESCRIPTION:
Inflammatory bowel disease (IBD) is comprised of two major disorders: ulcerative colitis (UC) and Crohn's disease(CD).CD is an autoimmune condition resulting in chronic gut inflammation that can be complicated by intestinal fibrosis and stricture formation. Ulcerative colitis is characterized by recurring episodes of inflammation limited to the mucosal layer of the colon. It commonly involves the rectum and may extend in a proximal and continuous fashion to involve other parts of the colon. Studies identified FAP to be overexpressed in uninflamed strictures compared with nonstrictured colonic regions in biopsies taken from Crohn's disease patients. But preliminary studies showed FAP was not overexpressed in colonic biopsies taken from healthy individuals or individuals with ulcerative colitis.68Ga-FAPI has been developed as a tumor-targeting agent as fibroblast activation protein is overexpressed in cancer-associated fibroblasts and inflammation. Recently we have published an article of the application of 68Ga-FAPI in IgG4-related disease which showed it was more sensitive than FDG in detecting a certain type of inflammations. Thus this prospective study is going to investigate whether 68Ga-FAPI PET/CT may be superior for diagnosis, therapy response assessment and follow-up of IBD than 18F-FDG PET/CT.

ELIGIBILITY:
Inclusion Criteria:

* suspected or confirmed untreated inflammatory bowel disease patients;
* 18F-FDG PET/CT within two weeks;
* signed written consent.

Exclusion Criteria:

* pregnancy;
* breastfeeding;
* known allergy against FAPI
* any medical condition that in the opinion of the investigator may significantly interfere with study compliance.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-08-01 (Actual); Primary Completion 2022-01-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Diagnostic value | through study completion, an average of 1 year
  Sensitivity and Specificity of 68Ga-FAPI PET/CT for inflammatory bowel disease in comparison with 18F-FDG PET/CT

SECONDARY OUTCOMES:
Metabolic parameters | through study completion, an average of 1 year
  Total Lesion Glycolysis (TLG) of bowel lesions are measured on 68Ga-FAPI PET/CT.
FAPI expression and SUV | through study completion, an average of 1 year
  Correlation between FAPI expression and SUV in PET
Disease burden assessement | through study completion, an average of 1 year
  Correlation between Total Lesion Glycolysis (TLG) of bowel lesions assessed on 68Ga-FAPI PET/CT and clinical parameters for inflammatory bowel disease
therapy response | through study completion, an average of 1 year
  Decrease of Total Lesion Glycolysis (TLG) on 68Ga-FAPI PET/CT after therapy

CONTACTS AND LOCATIONS:
Overall Officials: Yaping Luo, MD, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Luo Y, Pan Q, Xu H, Zhang R, Li J, Li F. Active uptake of 68Ga-FAPI in Crohn's disease but not in ulcerative colitis. Eur J Nucl Med Mol Imaging. 2021 May;48(5):1682-1683. doi: 10.1007/s00259-020-05129-7. Epub 2020 Nov 27. No abstract available. PMID 33247327